CLINICAL TRIAL: NCT01686984
Title: Influence of Inspiratory Flow Pattern on Exchange of Carbon Dioxide in Humans Without Primary Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012/381
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2015-05-14 (Estimated); Status verified 2015-05

CONDITIONS: Pulmonary Gas Exchange; Carbon Dioxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Altered breath (Experimental): The group where the investigators alter the inspiratory and expiratory aspects of a ventilated breath.
  Interventions: Other: Altered breath

INTERVENTIONS:
Other: Altered breath

SUMMARY:
The purpose of this study is to investigate how inspiratory flow pattern influences CO2 elimination in people without primary lung disease.

The hypothesis is that a long mean distribution time, caused by a long postinspiratory pause and high end-inspiratory flow, will promote CO2 exchange in the alveoli.

ELIGIBILITY:
Inclusion Criteria:

* No known primary lung disease

Exclusion Criteria:

* Primary lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2012-09; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Carbon dioxide elimination in a ventilator assisted breath. | 30 minutes

SECONDARY OUTCOMES:
Blood CO2 concentration. | 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Mikael Bodelsson, Professor, Principal Investigator — Division of Anesthesia, Skane University Hospital, Lund, Sweden
Locations (1):
- Division of Brain, Heart and Lungs, Neurosurgical Clinic, Skane University Hospital, Lund, Lund, Skåne County, Sweden

REFERENCES:
- [Derived] Sturesson LW, Malmkvist G, Allvin S, Collryd M, Bodelsson M, Jonson B. An appropriate inspiratory flow pattern can enhance CO2 exchange, facilitating protective ventilation of healthy lungs. Br J Anaesth. 2016 Aug;117(2):243-9. doi: 10.1093/bja/aew194. PMID 27440637